CLINICAL TRIAL: NCT05019781
Title: The Effectiveness of Kinesio Taping on Playing-related Pain, Function and Muscle Strength in Violin Players: a Randomized Controlled Clinical Trial
Brief Title: The Effectiveness of Kinesio Taping in Violin Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15082021
Record Dates: First submitted 2021-08-15; First posted 2021-08-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2021-08

CONDITIONS: Pain, Neck; Pain, Joint; Pain, Shoulder; Occupational Diseases; Musculoskeletal Pain
MeSH Terms: conditions — Neck Pain; Arthralgia; Shoulder Pain; Occupational Diseases; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- KT group (Experimental): Participants were received single session therapeutic tape application for one week.
  Interventions: Other: Therapeutic tape
- Placebo group (Placebo Comparator): Participants were received single session placebo tape application for one week.
  Interventions: Other: Placebo tape
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Other: Therapeutic tape — Tape was applied to sternocleidomastoid, upper trapezius, deltoid, flexor palmaris longus muscles as suggested by Kase et al. (Kase, Wallis, Kase, & Association, 2003). The tape was applied to the left side of the participants while sitting position because the violin is traditionally played by placing it on the left shoulder, balancing the neck using the left hand, and bowing with the right arm.
  Arms: KT group
Other: Placebo tape — The placebo tape was applied transverse to the muscle groups in two levels (a point of 10 cm above to wrist and elbow) with no tension when the participants were sitting position with the shoulder flexed at 90°, and the elbow flexed at 90°.
  Arms: Placebo group

SUMMARY:
This study aimed to investigate the effectiveness of Kinesio taping (KT) on playing-related pain, upper extremity and hand function, grip and pinch strength in violin players. One hundred seventeen participants who were professional violinists for at least two years were randomized to receive either therapeutic tape application (KT group), a sham tape application (placebo group) or no application (control group) for one week. The primary outcome was the Disabilities of the Arm, Shoulder and Hand (DASH) in one week. The secondary outcomes were the Visual Analogue Scale (VAS), the Purdue Pegboard Test, grip and pinch strength. Outcome measures were performed at baseline, immediately after the intervention, and one week later (follow-up). Participants were asked to play the "Violin Concerto No.2, Op.35", and pre-and post-performance pain and grip and pinch strength were assessed.

DETAILED DESCRIPTION:
Kinesio tape (KT), an alternative taping technique, is a method consisting of a tape with elastic properties and stretching capabilities used to treat pain or prevent injuries in conjunction with exercise.It has been concluded that KT intervention might not be helpful to reduce dystonic patterns or improve playing ability in musicians with focal hand dystonia. However, there is no enough study to conclude the effectiveness of KT application in Playing-related musculoskeletal disorders. Therefore, this study aimed to investigate the effect of KT on playing-related pain, upper extremity and hand function, grip and pinch strength in violin players compared to placebo KT application and control. As a secondary outcome, the investigators explored whether the pre-and post-performance effect of the KT on playing-related pain and grip and pinch strength.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 35 years;
2. professionally playing violin at least for two years;
3. having playing-related musculoskeletal pain at neck and upper extremity [Visual Analogue Scale (VAS) ≥3]
4. ability to read and write in Turkish; and
5. able to follow simple instructions.

Exclusion Criteria:

1. having significant musculoskeletal, neurologic, or cardiovascular disorders;
2. a history of surgery on the upper limbs in the previous six months;
3. the initiation of any analgesic intervention for musculoskeletal pain within the previous six weeks;
4. known allergies to tape; and
5. participation in physiotherapy and rehabilitation program in the last six months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Upper extremity function | Baseline
  The Disabilities of the Arm, Shoulder and Hand score is a self-administered questionnaire designed to evaluate single or multiple disorders and impairment levels in the upper limbs. It comprises 30 core questions and optional eight questions, which are scored on a 5-point Likert scale (no difficulty - unable). The cumulative score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.

SECONDARY OUTCOMES:
Upper extremity function | Follow-up (one week later)
  The Disabilities of the Arm, Shoulder and Hand score is a self-administered questionnaire designed to evaluate single or multiple disorders and impairment levels in the upper limbs. It comprises 30 core questions and optional eight questions, which are scored on a 5-point Likert scale (no difficulty - unable). The cumulative score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.
Playing-related pain | Baseline
  Playing-related pain was measured using the Visual Analogue Scale (VAS). The participants were asked to indicate their perceived pain while playing the violin on the 10 cm line between no pain and terrible pain. The score was determined by measuring the distance on a 10 cm line using a ruler.
Playing-related pain | Immediately after the intervention
  Playing-related pain was measured using the Visual Analogue Scale (VAS). The participants were asked to indicate their perceived pain while playing the violin on the 10 cm line between no pain and terrible pain. The score was determined by measuring the distance on a 10 cm line using a ruler.
Playing-related pain | Follow-up (one week later)
  Playing-related pain was measured using the Visual Analogue Scale (VAS). The participants were asked to indicate their perceived pain while playing the violin on the 10 cm line between no pain and terrible pain. The score was determined by measuring the distance on a 10 cm line using a ruler.
Playing-related pain | After one-week intervention (before playing Violin Concerto No.2, Op.35)
  Playing-related pain was measured using the Visual Analogue Scale (VAS). The participants were asked to indicate their perceived pain while playing the violin on the 10 cm line between no pain and terrible pain. The score was determined by measuring the distance on a 10 cm line using a ruler.
Playing-related pain | After one-week intervention (after playing Violin Concerto No.2, Op.35)
  Playing-related pain was measured using the Visual Analogue Scale (VAS). The participants were asked to indicate their perceived pain while playing the violin on the 10 cm line between no pain and terrible pain. The score was determined by measuring the distance on a 10 cm line using a ruler.
Hand function | Baseline
  The Purdue Pegboard Test was used to measure manual dexterity of both dominant and non-dominant hands. Participants were asked to place a pin in a vertical array of holes first with the right hand, then with the left hand, and following with both hands as quickly as possible in 30 s. In the final subtest, participants were asked to assemble a metal pin, washer, collar, and the second washer with both hands with the highest speed possible during 60 s.
Hand function | Immediately after the intervention
  The Purdue Pegboard Test was used to measure manual dexterity of both dominant and non-dominant hands. Participants were asked to place a pin in a vertical array of holes first with the right hand, then with the left hand, and following with both hands as quickly as possible in 30 s. In the final subtest, participants were asked to assemble a metal pin, washer, collar, and the second washer with both hands with the highest speed possible during 60 s.
Hand function | Follow-up (one week later)
  The Purdue Pegboard Test was used to measure manual dexterity of both dominant and non-dominant hands. Participants were asked to place a pin in a vertical array of holes first with the right hand, then with the left hand, and following with both hands as quickly as possible in 30 s. In the final subtest, participants were asked to assemble a metal pin, washer, collar, and the second washer with both hands with the highest speed possible during 60 s.
Hand function | After one-week intervention (before playing Violin Concerto No.2, Op.35)
  The Purdue Pegboard Test was used to measure manual dexterity of both dominant and non-dominant hands. Participants were asked to place a pin in a vertical array of holes first with the right hand, then with the left hand, and following with both hands as quickly as possible in 30 s. In the final subtest, participants were asked to assemble a metal pin, washer, collar, and the second washer with both hands with the highest speed possible during 60 s.
Hand function | After one-week intervention (after playing Violin Concerto No.2, Op.35)
  The Purdue Pegboard Test was used to measure manual dexterity of both dominant and non-dominant hands. Participants were asked to place a pin in a vertical array of holes first with the right hand, then with the left hand, and following with both hands as quickly as possible in 30 s. In the final subtest, participants were asked to assemble a metal pin, washer, collar, and the second washer with both hands with the highest speed possible during 60 s.
Grip and Pinch Strength | Baseline
  A hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer) is a practical tool to assess the hand's grip strength and pinch strength. For assessment of grip strength, the handle of the meter was adjusted at the second position. Each participant was instructed to squeeze the dynamometer's handle as hard as possible while positioning with the trunk upright; elbow flexed to 90°, forearm, and wrist in a neutral position. For assessment of pinch strength, the examiner held the distal end of the pinch gauge while the participant was instructed to squeeze the thumb pad according to different types of pinch grips (tip pinch, palmar pinch, key pinch). Assessments were repeated for the dominant and non-dominant hands. The mean values of the three grip strength and pinch strength measurements (kilogram-force) were calculated.
Grip and Pinch Strength | Immediately after the intervention
  A hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer) is a practical tool to assess the hand's grip strength and pinch strength. For assessment of grip strength, the handle of the meter was adjusted at the second position. Each participant was instructed to squeeze the dynamometer's handle as hard as possible while positioning with the trunk upright; elbow flexed to 90°, forearm, and wrist in a neutral position. For assessment of pinch strength, the examiner held the distal end of the pinch gauge while the participant was instructed to squeeze the thumb pad according to different types of pinch grips (tip pinch, palmar pinch, key pinch). Assessments were repeated for the dominant and non-dominant hands. The mean values of the three grip strength and pinch strength measurements (kilogram-force) were calculated.
Grip and Pinch Strength | Follow up (one week later)
  A hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer) is a practical tool to assess the hand's grip strength and pinch strength. For assessment of grip strength, the handle of the meter was adjusted at the second position. Each participant was instructed to squeeze the dynamometer's handle as hard as possible while positioning with the trunk upright; elbow flexed to 90°, forearm, and wrist in a neutral position. For assessment of pinch strength, the examiner held the distal end of the pinch gauge while the participant was instructed to squeeze the thumb pad according to different types of pinch grips (tip pinch, palmar pinch, key pinch). Assessments were repeated for the dominant and non-dominant hands. The mean values of the three grip strength and pinch strength measurements (kilogram-force) were calculated.
Grip and Pinch Strength | After one-week intervention (before playing Violin Concerto No.2, Op.35)
  A hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer) is a practical tool to assess the hand's grip strength and pinch strength. For assessment of grip strength, the handle of the meter was adjusted at the second position. Each participant was instructed to squeeze the dynamometer's handle as hard as possible while positioning with the trunk upright; elbow flexed to 90°, forearm, and wrist in a neutral position. For assessment of pinch strength, the examiner held the distal end of the pinch gauge while the participant was instructed to squeeze the thumb pad according to different types of pinch grips (tip pinch, palmar pinch, key pinch). Assessments were repeated for the dominant and non-dominant hands. The mean values of the three grip strength and pinch strength measurements (kilogram-force) were calculated.
Grip and Pinch Strength | After one-week intervention (after playing Violin Concerto No.2, Op.35)
  A hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer) is a practical tool to assess the hand's grip strength and pinch strength. For assessment of grip strength, the handle of the meter was adjusted at the second position. Each participant was instructed to squeeze the dynamometer's handle as hard as possible while positioning with the trunk upright; elbow flexed to 90°, forearm, and wrist in a neutral position. For assessment of pinch strength, the examiner held the distal end of the pinch gauge while the participant was instructed to squeeze the thumb pad according to different types of pinch grips (tip pinch, palmar pinch, key pinch). Assessments were repeated for the dominant and non-dominant hands. The mean values of the three grip strength and pinch strength measurements (kilogram-force) were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, PT, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No